CLINICAL TRIAL: NCT06016673
Title: Testing a Causal Model of Cognitive Control Deficits in Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Carter Bedford, Principal Investigator, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003574
Record Dates: First submitted 2023-08-23; First posted 2023-08-30 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: PTSD
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Each participant will receive stimulation to two brain areas (right dorsolateral prefrontal cortex and vertex) in a counterbalanced order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent theta burst stimulation to right dorsolateral prefrontal cortex (Experimental): Participants will receive intermittent theta burst stimulation (iTBS) to the experimental target area, the right dorsolateral prefrontal cortex (rDLPFC)
  Interventions: Procedure: Transcranial Magnetic Stimulation (TMS)
- Intermittent theta burst stimulation to vertex of the skull (Active Comparator): Participants will receive intermittent theta burst stimulation (iTBS) to the active comparator area, the vertex of the skull
  Interventions: Procedure: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation (TMS) — Participants will receive intermittent theta burst stimulation (iTBS) to two brain areas, the right dorsolateral prefrontal cortex (rDLPFC) and the vertex.

SUMMARY:
Testing a Causal Model of Cognitive Control Deficits in Posttraumatic Stress Disorder (PTSD)

DETAILED DESCRIPTION:
The purpose of the present study is to examine the effects of transcranial magnetic stimulation (TMS) on cognitive control among individuals with posttraumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Endorse lifetime exposure to at least one Criterion A traumatic event
* Report clinically significant posttraumatic stress disorder (PTSD) symptoms (score of ≥ 33 on the PTSD Checklist for DSM-5 [PCL-5]).

Exclusion Criteria:

* Endorse medical contraindication for neuromodulation (e.g., ferrous metal in head, seizure disorder, brain tumor, stroke, aneurysm, multiple sclerosis, etc.)
* Report an unstable medical condition or any current medical condition that precludes safe participation in the trial (e.g., unstable metabolic abnormality, unstable angina, etc.)
* Report any history or diagnosis of dementia or other cognitive disorder, which may interfere with engagement
* Report any history or diagnosis of Severe Traumatic Brain Injury
* Report any history or diagnosis of Schizophrenia, Schizoaffective Disorder, Delusional Disorder or other psychotic illness, which precludes safe participation in the trial
* Report a primary obsessive-compulsive disorder (OCD) diagnosis
* Report an active substance use disorder (within last 3 months) or any current substance use that precludes safe participation in the trial
* Report suicide risk that precludes safe participation in the trial, defined as clinical impression that the participant is at significant risk for suicide (i.e., greater than moderate level of suicide risk, in accordance with the Joiner et al. (1999) suicide risk framework)
* Report an inability to stop taking any medication that significantly lowers the seizure threshold (e.g., tricyclic antidepressants, clozapine, etc.)
* Report a current, planned, or suspected pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-02-03 (Actual)

PRIMARY OUTCOMES:
Performance on emotional working memory task | 5 hours
  Accuracy and reaction time on a task measuring working memory in the presence of trauma-related distractor images

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, PhD, Principal Investigator — Distinguished Research Professor
Locations (1):
- Florida State University College of Medicine, Tallahassee, Florida, United States